CLINICAL TRIAL: NCT02570464
Title: Aortic Cross-Clamping and Systemic Inflammatory Response in Humans: Effect of Ischemic Preconditioning
Acronym: CLARIS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: 2010/147/HP
Record Dates: First submitted 2015-10-02; First posted 2015-10-07 (Estimated); Last update posted 2016-05-12 (Estimated); Status verified 2016-05

CONDITIONS: Aortic Aneurysm
MeSH Terms: conditions — Aortic Aneurysm

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Patients undergoing aortic aneurysm surgery with RIPC (Experimental): Blood drawn is done for patient undergoing elective open infrarenal abdominal aortic aneurysm repair surgery with Remote ischemic preconditioning (RIPC)
  Interventions: Procedure: Remote ischemic preconditioning; Biological: Blood drawn
- Patients undergoing aortic aneurysm surgery without RIPC (Sham Comparator): Blood drawn is done for patient undergoing elective open infrarenal abdominal aortic aneurysm repair surgery without Remote ischemic preconditioning (RIPC)
  Interventions: Biological: Blood drawn

INTERVENTIONS:
Procedure: Remote ischemic preconditioning — Remote ischemic preconditioning is done for patients undergoing elective open infrarenal abdominal aortic aneurysm repair
  Arms: Patients undergoing aortic aneurysm surgery with RIPC
Biological: Blood drawn — Blood drawn is done for patients undergoing elective open infrarenal abdominal aortic aneurysm repair

SUMMARY:
Multiple organ dysfunction syndrome is a major cause of morbidity and mortality after abdominal aortic aneurysm (AAA) surgery. It is postulated that aortic cross-clamping during open AAA repair may cause ischemia-reperfusion (I/R) leading to the systemic releases of reactive oxygen species (ROS) and inflammatory cytokines which damage distant organs, including heart, kidney, and lung.

Ischemic preconditioning, first described in cardiac surgery, is a mechanism whereby tissues exposed to a brief period of nonlethal I/R develop resistance to subsequent ischemic insult. Remote ischemic preconditioning (RIPC), is a phenomenon whereby brief periods of ischemia followed by reperfusion in one organ (usually skeletal muscle) provide systemic protection from prolonged ischemia. The mechanisms through which RIPC confer organ protection remains unclear.

The hypothesis is that limb RIPC would reduce systemic inflammatory mediators produced by ischemia-reperfusion and thereby protect the remote organs.

A single-center, prospective, randomized, parallel-group controlled trial is conducted on patients undergoing elective open infrarenal AAA repair. Written informed consent is obtained from each participant. The study protocol was reviewed and approved by the Research Ethics Committee of Rouen, France.

Patients are divided in two groups : the sham-operated control group underwent surgery without RIPC and the RIPC group : Two cycles of intermittent crossclamping of the common iliac artery (right or left) with 10 minutes ischemia followed by 10 minutes reperfusion served as the RIPC stimulus, before prolonged ischemia.

Blood samples are collected for analysis at the following time points: before surgery (baseline), 1, 3 and 24 h after cross-clamp release (reperfusion). The systemic inflammatory response is measured using the serum concentrations of TNF-alpha, and IL 1, 4, 6, 10. Cardiac, renal and pulmonary functions are evaluated with usual biological markers and clinical monitoring until 28 days after surgery.

Aortic surgery is a perfect clinical model of ischemia-reperfusion which makes it possible to study the impact of RIPC in humans. This biological approach would help to better understand the mechanisms underlying this technique.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing elective open infrarenal abdominal aortic aneurysm repair
* Scheduled surgery
* Patients aged 30-85 years old

Exclusion Criteria:

* Patients undergoing endovascular treatment for infrarenal abdominal aortic aneurysm
* Patients younger than 30 years and older than 85 years
* pregnant women or nursing mother
* Adult under guardianship
* Refusal to sign a consent
* Patients whose survival at 28 days is unlikely
* Surgery requiring subphrenic aortic cross-clamping
* Emergency surgery
* Patients taking sulfonylureas or Nicorandil
* Patients having contraindication to clamp iliac arteries
* Dementia

Ages: 30 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2012-03; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Blood TNF-alpha rate | 24 hours post-surgery
  Blood TNF-alpha rate is measured after reperfusion

SECONDARY OUTCOMES:
Blood lactates rate | 24 hours post-surgery
  Blood lactates rate is measured after reperfusion
Blood I-CAM protein rate | 24 hours post-surgery
  Blood I-CAM protein rate is measured after reperfusion
Blood Interleukines 1 rate | 24 hours post-surgery
  Blood Interleukines 1 rate is measured after reperfusion
Blood Interleukines 4 rate | 24 hours post-surgery
Blood Interleukines 6 rate | 24 hours post-surgery
  Blood Interleukines 1 rate is measured after reperfusion
Blood Interleukines 10 rate | 24 hours post-surgery
  Blood Interleukines 10 rate is measured after reperfusion

CONTACTS AND LOCATIONS:
Overall Officials: Marie-Melody DUSSEAUX, MD, Principal Investigator — University Hospital, Rouen
Locations (1):
- Rouen University Hospital, Rouen, France

REFERENCES:
- [Derived] Liang F, Liu S, Liu G, Liu H, Wang Q, Song B, Yao L. Remote ischaemic preconditioning versus no remote ischaemic preconditioning for vascular and endovascular surgical procedures. Cochrane Database Syst Rev. 2023 Jan 16;1(1):CD008472. doi: 10.1002/14651858.CD008472.pub3. PMID 36645250